CLINICAL TRIAL: NCT03712020
Title: Investigating the Role of Active Versus Chronic Coronary Artery Calcification on Acute Myocardial Infarct: A Novel Pilot Study Using Sodium-Fluoride Positron Emission Tomography (PET) and Computed Tomography (CT) Techniques
Brief Title: Investigating the Role of Active Versus Chronic Coronary Artery Calcification on Acute Myocardial Infarct
Acronym: Active-AMI
Status: Completed | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/2183
Record Dates: First submitted 2016-05-31; First posted 2018-10-19 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigator aims to determine the feasibility of understanding the process of active versus chronic calcification using Na-F PET scan and contrast CT scan of the heart.

The patient cohort will consist of patients diagnosed to have either acute coronary syndrome (ACS) (comprising of either unstable angina pectoris or acute myocardial infarction) or suspected coronary artery disease (CAD). The PET images will be compared to images obtained from standard contrast CT of the coronaries. This study will provide additional insights about active versus non-active calcification amongst patients with ACS or suspected CAD.

DETAILED DESCRIPTION:
Contemporary techniques used to visualize coronary artery calcification include standard non-contrast computed tomography (CT) of the coronaries measuring amount of calcium deposition in the coronaries, contrast CT and more recently, using sodium-fluoride (Na-F) positron emission tomography (PET) to image coronary and valvular calcification. Na-F has been shown to accumulate in areas of active calcification where contrast CT of the heart has been shown to accumulate in areas of chronic calcification. The investigator aims to determine the feasibility of understanding the process of active versus chronic calcification using Na-F PET scan and contrast CT scan of the heart.

The patient cohort will consist of patients diagnosed to have either acute coronary syndrome (ACS) (comprising of either unstable angina pectoris or acute myocardial infarction) or suspected coronary artery disease (CAD). The PET images will be compared to images obtained from standard contrast CT of the coronaries. This study will provide additional insights about active versus non-active calcification amongst patients with ACS or suspected CAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of acute coronary syndrome
* Patients referred for workup of suspected coronary syndrome
* Able to provide written, informed consent.
* Age between (including) 50 years to 89 years old.

Exclusion Criteria:

* Pregnant & Lactating women
* weight <=180kg

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 patients
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Coronary artery calcification will be determined by Tc-99m MDP SPECT-CT and Na-F PET-CT | 12 months
  Na-F has been shown to accumulate in areas of active calcification where contrast CT of the heart has been shown to accumulate in areas of chronic calcification. We aim to determine the feasibility of understanding the process of active versus chronic calcification using Na-F PET scan and contrast CT scan of the heart.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Koh, Principal Investigator — National Heart Centre

IPD SHARING:
Plan to Share IPD: Undecided